CLINICAL TRIAL: NCT02722616
Title: Ultrasound System For Non-Invasive, Real-Time Monitoring of Abdominal Soft Tissue
Brief Title: Ultrasound Monitoring of Abdominal Soft Tissue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ultrasound vendor cannot support the study
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: J14176; IRB00053627 (Other: JHMIRB); R01CA161613 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2016-03-30 (Estimated); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer; Liver Cancer
Keywords: Ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pancreatic Cancer (Active Comparator): A 4D ultrasound scan of the pancreas will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the pancreas motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup can be reproduced during treatment delivery. The ultrasound probe in the CT image will be contoured and radiation beams that directly pass through the ultrasound probe will be avoided.
  On each treatment day, 4D ultrasound images will be acquired continuously during beam on time to monitor pancreas motion. Intra-fraction CBCT images acquired during treatment will be registered with reference CT images. Organ motion registered by ultrasound will be compared to motion recorded by CBCT and the accuracy of the ultrasound system will be evaluated.
  Interventions: Device: Ultrasound scan of the pancreas
- Liver Cancer (Active Comparator): A 4D ultrasound scan of the liver will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the liver motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup could be reproduced during treatment delivery.
  On each treatment day, 4D ultrasound images will be acquired continuously during beam on time to monitor liver motion. The system will record all relevant images, but will not be used in clinical decision making. Intra-fraction CBCT images acquired during treatment will be registered with reference CT images. Organ motion registered by ultrasound will be compared to motion recorded by CBCT and the accuracy of the ultrasound system will be evaluated.
  Interventions: Device: Ultrasound scan of the Liver
- Healthy Volunteer (Other): A reference ultrasound scan will be conducted on each subject during breath-hold. Subjects will be required to lie in supine position and engaged with ABC; an ultrasound probe will be placed at the abdomen area with minimal pressure applied. Continuous motion monitoring is achieved by acquiring 4D ultrasound images using a motorized 3D ultrasound probe to image the pancreas, liver and other intra-abdominal organs continuously. Several 4D ultrasound scans will be collected during subsequent breath-holds that serve as secondary images. Additional registration of ultrasound images will be performed with Velocity software to evaluate accuracy of automated registration software in the ultrasound system.
  Interventions: Drug: Reference ultrasound

INTERVENTIONS:
Device: Ultrasound scan of the pancreas — A 4D ultrasound scan will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the pancreas motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup can be reproduced during treatment delivery.
  Other Names: 4D ultrasound
  Arms: Pancreatic Cancer
Device: Ultrasound scan of the Liver — A 4D ultrasound scan will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the liver motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup could be reproduced during treatment delivery. The ultrasound probe in the CT image will be contoured and radiation beams that directly pass through the ultrasound probe will be avoided.
  Other Names: 4D ultrasound
  Arms: Liver Cancer
Drug: Reference ultrasound — A reference ultrasound scan will be conducted on each subject during breath-hold. Subjects will be required to lie in supine position and engaged with ABC; an ultrasound probe will be placed at the abdomen area with minimal pressure applied. Continuous motion monitoring is achieved by acquiring 4D ultrasound images using a motorized 3D ultrasound probe to image the pancreas, liver and other intra-abdominal organs continuously. Several 4D ultrasound scans will be collected during subsequent breath-holds that serve as secondary images.
  Other Names: 4D ultrasound
  Arms: Healthy Volunteer

SUMMARY:
This research study is being done to collect data and analyze the motion of soft tissue in the abdomen (liver, pancreas, stomach and intestines) of people who have pancreatic and liver cancer as well as healthy volunteers.

During the study researchers will look at the movement of organs in the abdomen that naturally occurs with breathing and with a bowel movement.

This study will examine the differences between abdominal soft tissue motion in healthy volunteers and in cancer patients with the goal of developing a better way to manage and minimize the abdominal soft tissue motion. Accurate location of the tumor is very important in treatment delivery and reduction of toxicity.

DETAILED DESCRIPTION:
Within the last decade, Linac based stereotactic body radiation therapy (SBRT) has been shown to be an effective treatment option for pancreas1, 2 and liver3, 4 tumors. SBRT delivers high doses of radiation therapy to the tumor over only 1-5 treatments. Because of the spatial precision of SBRT, it is feasible to administer a high radiation dose in only a few treatments. By minimizing the amount of radiation to surrounding healthy tissue, it is possible to decrease the rate of toxicity/complication and increase the radiation dose to cancerous tissue, thereby allowing better local control.

SBRT of the abdomen has been limited by the movement of intra-abdominal organs that naturally occurs with respiration and bowel movement. Organ motion occurs both intra- and inter-fractionally. While intra-fractional motion is a result of respiration, peristalsis and cardiac motion, the magnitude of inter-fractional target motion is dependent of daily variations in organ filling, weight change, tumor growth and radiation induced changes of tissue. Tumor movement may lead to tumor displacement and suboptimal dose delivery. Accurate localization of the target is very important to improve treatment delivery accuracy and reduce toxicity of the treatment. To evaluate tumor motion due to breathing motion, a four dimensional (4D) CT simulation scan is performed. If the tumor moves more than 3 mm during a breathing cycle, breathing motion management is employed using Active Breathing Control (ABC) technique. ABC requires the patient to hold his/her breath within the proper tidal volume while treatment is delivered, while free breathing may be resumed between periods of treatment. This technique limits the delivery of RT to specific phases of the respiratory cycle so as to minimize the influence of breathing on the delineated tumor.

Despite significant progress made in ABC technique, tumor and organ motion could only be minimized and not eliminated completely with this technique. Assessing patient specific tumor/organ motion (both intra- and interfractional) throughout the course of SBRT treatment offers the possibility of ensuring delivery of the prescribed target dose while simultaneously minimizing normal tissue damage. In order to monitor the abdominal soft tissue motion, the Department of Radiation Oncology has developed a 4D ultrasound technique based on an ultrasound probe holder and a continuous motion monitoring software. The 4D ultrasound image is acquired by using a motorized 3D ultrasound probe and image continuously. 4D ultrasound is a new non-ionizing and non-invasive imaging technique that continuously monitors the tumor motion during the radiation treatment in real time.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1: Healthy adult (age >18 years)
* Arm 2: Pancreatic cancer patients (age >18 years) currently receive SBRT treatment at Johns Hopkins University (JHU)
* Arm 3: Hepatic cancer patients (age >18 years) currently receive SBRT treatment at JHU

Exclusion Criteria:

* Children (age < 18 years) are excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pancreatic Cancer: A 4D ultrasound scan of the pancreas will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the pancreas motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup can be reproduced during treatment delivery. The ultrasound probe in the CT image will be contoured and radiation beams that directly pass through the ultrasound probe will be avoided.
  On each treatment day, 4D ultrasound images will be acquired continuously during beam on time to monitor pancreas motion. Intra-fraction CBCT images acquired during treatment will be registered with reference CT images. Organ motion registered by ultrasound will be compared to motion recorded by CBCT and the accuracy of the ultrasound system will be evaluated.
  Ultrasound scan of the pancreas: A 4D ultrasound scan will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the pancreas motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup can be reproduced during treatment delivery.
- Liver Cancer: A 4D ultrasound scan of the liver will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the liver motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup could be reproduced during treatment delivery.
  On each treatment day, 4D ultrasound images will be acquired continuously during beam on time to monitor liver motion. The system will record all relevant images, but will not be used in clinical decision making. Intra-fraction CBCT images acquired during treatment will be registered with reference CT images. Organ motion registered by ultrasound will be compared to motion recorded by CBCT and the accuracy of the ultrasound system will be evaluated.
  Ultrasound scan of the Liver: A 4D ultrasound scan will be acquired at the time at simulation and used as a reference ultrasound image for localizing tracking target. The ultrasound probe will be placed at the abdominal area to monitor the liver motion. The probe will remain in place during the CT scan. Patient setup and the ultrasound probe location will be recorded so that the same setup could be reproduced during treatment delivery. The ultrasound probe in the CT image will be contoured and radiation beams that directly pass through the ultrasound probe will be avoided.
Period: Overall Study
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer
Started | 2 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Sponsor closed study after one month | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sponsor closed study after 2 patients in Pancreatic Cancer arm of the study were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 76 [74 to 78] |  |  | 76 [74 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 1 |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 0 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Soft-tissue Movement
Description: Measuring changes in abdominal soft-tissue movement through 4D ultrasound system
Time Frame: change in abdominal soft-tissue movement from baseline to 3 weeks
Population: Patients were consented, enrolled and taken off study during the period 5/3/2016-6/9/2016. Data was not collected or analyzed because the sponsor closed the study early. In order to collect and analyze the data, treatment would have to have been completed.
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Tissue Change During Radiation Treatment
Description: monitoring of tumor and surrounding organ/tissue during pancreas and liver SBRT treatments using 4D ultrasound system
Time Frame: change in tumor tissue from baseline to 3 weeks
Population: as for outcome 1
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Change 4D Ultrasound to Traditional Cone-beam Computed Tomography (CBCT) Monitoring
Description: Evaluate accuracy of the 4D ultrasound motion monitoring system compare to CBCT based intra-fraction motion monitoring during pancreas and liver SBRT treatments
Time Frame: change in imaging studies of 4D ultrasound from baseline to 3 weeks
Population: as for outcome 1
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Dosimetry Measurements
Description: Evaluation of dosimetry differences due to target/organ motion observed
Time Frame: dosimetric changes in abdominal soft-tissue movement from baseline to the end of radiation treatment at 3 weeks
Population: as for outcome 1
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not collected
Arm/Group | Pancreatic Cancer | Liver Cancer | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT02722616/Prot_SAP_000.pdf